CLINICAL TRIAL: NCT02284126
Title: Topical Vancomycin for the Reduction of Surgical Site Infections in Neurosurgery
Brief Title: Topical Vancomycin for Neurosurgery Wound Prophylaxis
Acronym: Vanguard
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Cornell University (Other); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, E. Sander Connolly, Bennett M. Stein Professor of Neurological Surgery Vice Chairman of Neurosurgery Director, Cerebrovascular Research Laboratory Surgical Director, Neuro-Intensive Care Unit, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AAAN3703; 1R01HS022903-01 (AHRQ)
Record Dates: First submitted 2014-11-03; First posted 2014-11-05 (Estimated); Results first posted 2021-01-25 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-09

CONDITIONS: Infection; Surgery; Nervous System Diseases
Keywords: Vancomycin; Anti-Infective Agents, Local; Craniotomy; Surgical Site Infection; Wound Prophylaxis; Anti-Bacterial Agents; Neurosurgical Procedures; Administration, Topical; Antibiotic Prophylaxis; Antibiotics; Prophylaxis; Neurosurgery; Bacterial Infections; Central Nervous System Infections
MeSH Terms: conditions — Infections; Nervous System Diseases; Surgical Wound Infection; Bacterial Infections; Central Nervous System Infections | interventions — Vancomycin; Injections

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Topical Vancomycin (Experimental): Treatment group, receive 2 g topical vancomycin hydrochloride (1 g applied as powder, 1 g mixed with sterile solution and applied as paste) at the time of closure, in addition to the standard of care for wound prophylaxis
  Interventions: Drug: Vancomycin
- Standard of Care (No Intervention): Control group, receive standard of care only

INTERVENTIONS:
Drug: Vancomycin — Topically applied powder and paste to surgical site at time of closure.
  Other Names: Vancomycin Hydrochloride for Injection
  Arms: Topical Vancomycin

SUMMARY:
This study is a collaboration between New York Presbyterian (NYP)-Columbia and NYP-Cornell that seeks to evaluate the use of topical vancomycin and its reduction on surgical site infection (SSI) in neurosurgical procedures. Adult patients undergoing neurosurgery at either institution will be eligible for participation in this randomized control trial. Patients randomized to the treatment group will receive 2g of vancomycin applied as a powder or paste to the wound site and/or bone flap. Subjects in the control group will receive the current standard of care without topical vancomycin. All subjects will undergo swabbing of the anterior nares and the surgical site prior to surgery, once 10-14 days following the operation and 90 days following the operation. The primary outcome measure will be surgical site infection, assessed daily throughout the hospital stay, at the first follow-up visit, and by telephone at 14-30 days and 90 days (+/- 7 days). Secondary outcomes will include length of hospital stay, length of intensive care stay, rate of reoperation and patient mortality. In addition, systemic vancomycin levels will be assessed at 6 hours and 20 hours postoperatively in each patient. Patients who have an external ventricular drain in place will have vancomycin levels assessed daily. In patients who have cranial drains placed, vancomycin concentrations will be analyzed from daily in wound drainage. Skin and nasal flora will be analyzed to assess the impact of topical vancomycin on the patient microbiome. Although there has been a decrease in the incidence of infections following craniotomy secondary to prophylactic intravenous antibiotics, proper sterile techniques, and other interventions, SSIs continue to significantly impact morbidity, mortality, and cost burden. Although never studied in neurosurgical procedures other than instrumented spine, the application of topical vancomycin to the surgical site prior to wound closure has demonstrated a reduction in SSIs in spine, cardiac and ophthalmologic procedures. The benefits of using prophylactic vancomycin topically, as opposed to intravenously, include reduced systemic levels of the drug, and therefore, a decreased probability of adverse events related to the drug, such as inducing resistance among the native flora. The investigators propose a single-blinded randomized control trial to evaluate the effectiveness of topical vancomycin in reducing SSIs rates following neurosurgical procedures.

DETAILED DESCRIPTION:
Surgical-site infections (SSIs) occur in up to 500,000 patients per year in the United States. Patients with SSIs require significantly longer hospital stays and higher health care expenditures. In fact, it is estimated that SSIs are responsible for almost 4 million excess hospital days and billions of dollars in added hospital charges every year. Additionally, SSIs are a significant source of morbidity and mortality for surgical patients. Thus, prompt and definitive measures are necessary in order to redress this significant public health concern. Over the past few decades, the implementation of a number of preventative measures-including improved techniques in pre-operative skin antisepsis and antibiotic prophylaxis-have led to significant reductions in the rate of SSIs. Studies have demonstrated that approximately half of all SSIs are preventable with the proper use of prophylactic antibiotics. Despite these dramatic improvements, SSIs remain a tremendous burden on the healthcare system. Our unpublished analysis of the National Inpatient Sample (NIS) in 2010 identified 117,000 craniotomies with a 2.4% rate of infection and 1.37% rate of Methicillin-resistant Staphylococcus aureus (MRSA)-associated infection. Extrapolating to the full national population, there were 585,000 craniotomies and 14,040 post-operative infections. Published series report the rate of infection in intracranial neurosurgery to range from 1% to as high as 11%. This rate varies depending on the presence of hardware, prior radiotherapy, procedure duration, re-operation, and the presence of a CSF leak. The 30-day outcome associated with SSI following craniotomy was recently reported to be a minor disability in 12.8%, major disability in 7.7% and death in 5.1%. The financial burden of nosocomial infection in neurosurgery makes up a disproportionate component of the total national cost burden. A study of nosocomial infection in the US in 1995 estimated a per-patient cost of $2100 and a total cost of $4.5 billion while a recent British study focusing on post-craniotomy SSI identified a per-SSI cost of £9283, or $14,166. Given the tremendous potential for lifelong morbidity and mortality as a result of cranial SSIs, further reductions in the rate of SSI would be essential for the benefit of neurosurgical patients, as well as for the healthcare system as a whole.Topical formulations of vancomycin offer the possibility of direct application to the surgical wound, with minimal additional systemic drug exposure. Adjunctive vancomycin powder applied topically to surgical wound edges has been shown to significantly lower the SSI rate in both cardiothoracic surgery and spinal surgery. Importantly, laboratory analyses of blood and wound drainage samples from patients treated with vancomycin powder have demonstrated high vancomycin concentrations in the surgical wound, and simultaneously low drug concentrations in the peripheral blood, thereby confirming minimal systemic absorption in the setting of enhanced protection of the surgical site. Furthermore, there have been no reports of an increased rate of drug-related complications with the addition of vancomycin powder to standard antibiotic prophylaxis regimens.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18+) neurosurgical procedure (ie.Craniotomy, Craniectomy, and Cranioplasty)

Exclusion Criteria:

* Creatinine > 1.50 mg/dL on admission
* Vancomycin allergy (documented or self-reported)
* Evidence of infection at or near the planned surgical site
* No planned dural or dural-substitute closure
* Spinal instrumentation (topical vancomycin is already standard of care)
* No surface area to apply:Carotid endarterectomy, MRI-guided laser ablation
* Trans-sphenoidal approach
* Acoustic neuroma resection
* Surgeon preference for or against use in the given procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1103 (Actual)
Dates: Start 2014-10; Primary Completion 2019-11 (Actual); Study Completion 2020-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E. Sander Connolly, M.D., Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Radwanski RE, Christophe BR, Pucci JU, Martinez MA, Rothbaum M, Bagiella E, Lowy FD, Knopman J, Connolly ES. Topical vancomycin for neurosurgery wound prophylaxis: an interim report of a randomized clinical trial on drug safety in a diverse neurosurgical population. J Neurosurg. 2018 Dec 14;131(6):1966-1973. doi: 10.3171/2018.6.JNS172500. Print 2019 Dec 1. PMID 30554184

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Topical Vancomycin | Standard of Care
Started | 552 | 551
Completed | 484 | 489
Not Completed | 68 | 62

BASELINE CHARACTERISTICS:
Population: Out of 1103 enrolled subjects, only 973 subjects completed the study and their data have been analyzed and presented here.
Groups:
- Total: Total of all reporting groups
Arm/Group | Topical Vancomycin | Standard of Care | Total
Number analyzed (Participants) | 484 | 489 | 973
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (16.1) | 53.3 (17.0) | 53.7 (16.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 276 | 280 | 556
  Male | 208 | 209 | 417
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 50 | 43 | 93
  Not Hispanic or Latino | 403 | 403 | 806
  Unknown or Not Reported | 31 | 43 | 74
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 19 | 24 | 43
  Native Hawaiian or Other Pacific Islander | 3 | 1 | 4
  Black or African American | 39 | 33 | 72
  White | 337 | 339 | 676
  More than one race | 18 | 18 | 36
  Unknown or Not Reported | 67 | 73 | 140

OUTCOME MEASURES:

1. Primary Outcome: Any Surgical-site Infection as Evidenced by Surgeon or Attending Physician Diagnosis, or Signs and Symptoms of Infection Assessed by Phone Call Interview or at In-office Follow-up Consultation
Description: Classified as superficial incisional, deep incisional, or organ/space (intradural) infection
Time Frame: 30 days & 90 days (+/- 7 days) postoperatively
Measure: Number; unit: participants
Arm/Group | Topical Vancomycin | Standard of Care
Number analyzed (Participants) | 484 | 489
participants
  Subject visited doctor and received antibiotics | 18 | 19
  Subject reports any possible symptom of surgical site infection | 344 | 355
  Positive skin culture or hospital readmission for surgical site infection | 5 | 4

2. Primary Outcome: Number of Subjects That Reported Any Surgical-site Infections
Description: As evidenced by surgeon or attending physician diagnosis, or signs and symptoms of infection assessed by phone call interview or at in-office follow-up consultation. Classified as superficial incisional, deep incisional, or organ/space (intradural) infection.
Time Frame: 30 days & 90 days (+/- 7 days) postoperatively
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Topical Vancomycin | Standard of Care
Number analyzed (Participants) | 484 | 489
participants | 344 | 355

3. Secondary Outcome: Number of Participants With Positive Serum Vancomycin Levels
Description: Vancomycin levels in serum will be tested after surgery, any additional fluid collections, but if and only if clinically indicated. A serum vancomycin level of >3.0 mg/dl is considered positive.
Time Frame: 6-20 hours post-operatively
Population: 440 participants who were administered vancomycin provided serum samples for analysis. The remaining participants were discharged on the same day as their operation and thus were not available to provide serum samples.
  Serum samples were not collected from participants who received standard of care.
Measure: Count of Participants; unit: Participants
Arm/Group | Topical Vancomycin | Standard of Care
Number analyzed (Participants) | 440 | 0
Participants | 21 |

4. Secondary Outcome: Number of Participants Who Developed a Previously Undetected Vancomycin Resistance
Description: Microbial swabs will be obtained by the clinical coordinator preoperatively, post-operatively, at 10-14 days and at 90 days. Staph aureus isolates from mannitol growth will be tested for vancomycin resistance.
Time Frame: 90 days postoperatively
Population: Swabs were collected only from participants who received Vancomycin.
Measure: Count of Participants; unit: Participants
Arm/Group | Topical Vancomycin | Standard of Care
Number analyzed (Participants) | 484 | 0
Participants | 0 |

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Topical Vancomycin | Standard of Care
All-Cause Mortality (participants affected / at risk) | 5/552 | 6/551
Serious Adverse Events (participants affected / at risk) | 49/552 | 65/551
Other Adverse Events (participants affected / at risk) | 121/552 | 119/551
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topical Vancomycin (N=552) | Standard of Care (N=551)
Hearing loss (Ear and labyrinth disorders) | 4 (4) | 7 (7)
Death (General disorders) | 5 (5) | 6 (6)
Allergy Symptoms (Immune system disorders) | 0 (0) | 1 (1)
Gastrointestinal Changes (Gastrointestinal disorders) | 1 (1) | 0 (0) — E. Coli
Surgical Site Infection (Infections and infestations) | 4 (4) | 4 (4)
Unplanned Medical Visit (General disorders) | 21 (22) | 37 (37)
Urinary Tract Infeciton (Infections and infestations) | 1 (1) | 3 (3)
Aspiration Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 3 (3) | 1 (1)
Vision Impairment (Nervous system disorders) | 1 (1) | 2 (2)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Pancreatic Necrosis (Endocrine disorders) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 1 (1) | 1 (1)
Bleeding at drain site (General disorders) | 0 (0) | 1 (1)
Left Ventricular Thrombus (Cardiac disorders) | 0 (0) | 1 (1)
Facial Sensory Loss (Nervous system disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Meningitis (Nervous system disorders) | 1 (1) | 1 (1)
Dysarthria/Dysphagia (Nervous system disorders) | 0 (0) | 3 (3)
Hemiparesis (Nervous system disorders) | 1 (1) | 3 (3)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Cognitive Impairment (Nervous system disorders) | 2 (2) | 2 (2)
Stroke/Cerebrovasular accident (Nervous system disorders) | 3 (3) | 2 (2)
Gait instability (General disorders) | 0 (0) | 1 (1)
Drop foot (Nervous system disorders) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 0 (0)
Pulmonary Embolism (Vascular disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Pneumocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Epidural Abscess (General disorders) | 1 (1) | 0 (0)
Discharge (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topical Vancomycin (N=552) | Standard of Care (N=551)
Allergy Symptoms (Immune system disorders) | 32 (32) | 33 (33)
Gastrointestinal changes (Metabolism and nutrition disorders) | 30 (33) | 34 (36) — Diarrhea, nausea, constipation, vomiting, etc
Hearing Change (Ear and labyrinth disorders) | 24 (26) | 26 (27)
Unplanned Medical Visit (General disorders) | 35 (38) | 26 (30)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-23): https://cdn.clinicaltrials.gov/large-docs/26/NCT02284126/Prot_SAP_000.pdf